CLINICAL TRIAL: NCT05532566
Title: Quercus Ilex and Quercus Robur Allergen Extracts. Determination of the in Vivo Allergenic Potency in Histamine Equivalent Units (HEP).
Brief Title: Quercus Ilex and Quercus Robur Allergen Extracts Standardisation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: T525-STD-043; 2020-005388-30 (EudraCT Number)
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-05

CONDITIONS: Allergic Reaction; Allergic Skin Reaction; Allergy Pollen
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic, Seasonal | interventions — grass pollen extract, alum-adsorbed

STUDY DESIGN:
Intervention Model Description: Phase II, open-label, non-randomized trial, with no control group of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extract Q. ilex + extract Q. robur + positive control + negative control (Experimental): There is only one treatment arm. In each subject, one drop of each of the 3 concentrations of each allergenic extract (2 extracts) will be applied in addition to the positive control (histamine 10mg/mL) and the negative control, with prick test.
  Quercus ilex: 2,500, 500 and 100 μg/mL Quercus robur: 2,500, 500 and 100 μg/mL
  Interventions: Other: Allergenic extract

INTERVENTIONS:
Other: Allergenic extract — In each subject a drop of each of the 3 concentrations of both allergenic extracts will be applied in addition to the positive control (histamine) and the negative control. The application will be made in duplicate on the anterior face of the subject's arm. The distance between each application should be approximately 4 cm.
  Other Names: Allergenic Quercus ilex and Quercus robur extract

SUMMARY:
The objective of this study is to determine the biological activity of Quercus illex and Quercus robur allergen extracts in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
The trial will consist of a single visit, in which the following procedures will be carried out:

* Demographic data.
* Clinical history.
* Inclusion/exclusion criteria.
* General examination.
* Performance of prick-tests (3 concentrations of Quercus ilex allergenic extract, 3 concentrations of Quercus robur allergenic extract, positive control and negative control).
* Obtaining a blood sample from the patient to create a pool of sera for the "in vitro" standardization of the allergenic extract. This pool of sera is necessary for the characterization of the Company's standard. Each serum sample will be stored in a tube that will be labeled with the subject number and frozen. These serum samples will remain in the freezer until the study is completed. When the study is completed, they will be transported to the laboratory, where all sera will be pooled. This "pool" of sera will be used to perform the complementary in vitro standardization tests. These include ELISA for measurement of inhibition against specific IgE, etc. These serum samples are not destroyed. They are pooled together to form a pool that will be used, as described in the previous paragraph, in all the in vitro tests necessary to standardize and characterize this extract and produce its corresponding HIRP (In-house reference preparation), as indicated by the Royal Spanish Pharmacopoeia and the European Pharmacopoeia. This pool of sera is not destroyed, it is used in the in vitro analyses necessary for the standardization of new batches of this allergenic extract. Once the pool has been formed, the tubes containing the original serum samples are destroyed.
* Evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must live in a geographical area where allergic problems caused by Quercus ilex and Quercus robur are relevant.
* Positive clinical history of inhalant allergy (rhinitis and/or rhinoconjunctivitis and/or asthma) to asthma) to Quercus ilex and Quercus robur.
* A positive prick-test (mean papule diameter ≥ 3 mm) with an extract of the same allergen and/or presence of specific IgE against that allergen.
* The mean papule area obtained with Histamine dichlorhydrate at 10 mg/mL should be ≥ 7 mm2.
* Age: Between 18 and 64 years old.
* Subjects must be able to give informed consent.

Exclusion Criteria:

* Subjects should not be excluded in terms of low or high sensitivity to Quercus ilex and Quercus robur.
* Subjects outside the age range.
* Subjects who have previously received immunotherapy in the last 5 years for the treatment of asthma or rhinoconjunctivitis for the treatment of asthma or allergic rhinoconjunctivitis induced by allergens that may interfere with Quercus ilex and Quercus robur extracts.
* Subjects with significant symptoms of rhinoconjunctivitis and/or bronchial asthma in which the suspension of the systemic antihistamine treatment is contraindicated.
* Subjects who have previously presented a severe secondary reaction during the performance of diagnostic skin tests by prick test.
* Subjects under treatment with ß-blockers.
* Subjects clinically unstable (acute asthma, febrile, etc.).
* Subjects with active urticaria lesions, severe active dermographism, severe atopic dermatitis, sunburn, eczema, psoriasis lesions in the area where the prick test is performed (risk of false positives).
* Subjects with active viral infection by herpes simplex or herpes varicella zoster in the area where the prick test is performed.
* Subjects with any pathology in which the administration of adrenaline is contraindicated (hyperthyroidism, HTA, cardiopathy, etc.).
* States of the subject in which he/she cannot offer cooperation and severe psychiatric disorders.
* Pregnant women or women at risk of pregnancy and lactating women.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Size of the induced papule on the skin | 15 minutes
  Size of the induced papule on the skin when applying each of the concentrations of the allergenic extracts and the positive (histamine) and negative controls, using the prick test.
Adverse reactions | 30 minutes
  Mild secondary reactions such as pruritus, erythema, local edema, etc. There is a risk, infrequent and exceptional, of systemic reactions, sometimes severe (urticaria, asthma, anaphylactic shock, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Subiza, MD, Principal Investigator — Clinica Subiza, centro de asma y alergia
Locations (1):
- Clínica Subiza, centro de asma y alergia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sjoholm I. Standardisation of allergens in Europe. Arb Paul Ehrlich Inst Bundesamt Sera Impfstoffe Frankf A M. 1997;(91):107-10. PMID 9383897
- [Background] Larsen JN, Dreborg S. Standardization of Allergen Extracts. Methods Mol Biol. 2019;2020:63-76. doi: 10.1007/978-1-4939-9591-2_5. PMID 31177492
- [Background] Arntzen FC. Progress in common Nordic Guidelines for the Registration of Allergen Preparations. Arb Paul Ehrlich Inst Georg Speyer Haus Ferdinand Blum Inst Frankf A M. 1983;(78):25-8. No abstract available. PMID 6625583